CLINICAL TRIAL: NCT07086365
Title: Feasibility of Using Immersive Virtual Functional Rehabilitation for Recovery of Upper Extremity Function in Patients With Early-stage Stroke: a Pilot Study
Acronym: IMVR Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Alemana de Santiago (Other)
Responsible Party: Principal Investigator, Margarita Venegas, Ricardo Vasquez, Clinica Alemana de Santiago
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 1134 UIEC
Record Dates: First submitted 2025-05-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Stroke Acute
Keywords: stroke; rehabilitation; neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Pilot study evaluating the feasibility of using an immersive virtual reality device in patients with stroke in the acute and sub-acute stages. Preliminary functional outcomes about upper extremity function are also assessed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 session (Other): Participants receive 10 sessions of intervention with virtual inmersive reality.
  Virtual reality with hand tracking and immersive environment
  Interventions: Device: Immersive virtual reality
- 20 sessions (Other): Participants receive 20 sessions of intervention with virtual inmersive reality. Virtual reality with hand tracking and immersive environment.
  Interventions: Device: Immersive virtual reality

INTERVENTIONS:
Device: Immersive virtual reality — Virtual reality with hand tracking and immersive environment
Device: Immersive Virtual Reality — Immersive virtual reality is a digital therapeutic approach to enhance neuroplasticity using virtual environment and hand tracking for functional motion in upper extremity
  Other Names: Extended reality.; Digital therapeutics.

SUMMARY:
Feasibility of using immersive virtual functional rehabilitation for recovery of upper extremity function in patients with early-stage stroke: a pilot study

DETAILED DESCRIPTION:
Background: Immersive virtual reality (IVR)-based rehabilitation provides high-intensity, engaging, task-oriented training and motor exploration for upper limb (UL) recovery post-stroke. However, its feasibility and dose-response effects remain unclear.

Objective: To evaluate the feasibility and dose-response effects of IVR-based rehabilitation for UL recovery in early stroke patients.

Methods: A pilot trial included 12 early-stage stroke patients randomized into two groups: Group A (10 IVR sessions + conventional rehabilitation [CR]) and Group B (20 IVR sessions + CR). Feasibility outcomes included adherence, usability (User Satisfaction Evaluation Questionnaire [USEQ], System Usability Scale [SUS]), system operability, and adverse effects. Motor outcomes, categorized by the International Classification of Functioning, Disability, and Health (ICF), assessed UL impairment (Fugl-Meyer Assessment, Medical Research Council scale), activity (Box and Block Test), and participation (Motor Activity Log 30). Blinded therapists conducted assessments at baseline, post-intervention, and 4-week follow-up. Dose-response was analyzed using Probability of Superiority (PS).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* first episode of stroke (ischemic or hemorrhagic)
* time since stroke onset between 0 to 6 months
* upper limb motor impairment with the National Institutes of Health Stroke Scale arm motor sub-item score between 1 and 4
* medically stable parameters for rehabilitation initiation.

Exclusion Criteria:

* Delirium diagnosed using the Confusion Assessment Method
* Montreal Cognitive Assessment Scale <18
* Severe visual/perceptual deficits (spatial neglect affecting >70% of trials or visual acuity <20/200)
* previous participation in virtual reality-based rehabilitation
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
System Usability Scale [SUS] | The treatment providers fill out the questionnaire at the end of treatment. It depends of the group patient: 10 or 20-session treatment.
  Questionnaire completed by the handlers who administer the immersive virtual reality system
User Satisfaction Evaluation Questionnaire [USEQ] | Administered within the first 7 days of using the immersive virtual reality device
  Questionnaire of 5 questions with 5 options based on likert rate. Is filled for the patient recruited

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity | It is administered in three stages: Baseline or day 1 (pre treatment). In the week number 4 (post treatment). Up to 8 weeks (follow-up). Through study completion, an average of 6 months.
  Clinical assessment scale for upper extremity function. It evaluates various functional areas of the upper extremity: wrist, hand, coordination, and speed. This provides a total of 66 motor function points.
Motor Activity Log | It is administered in three stages: Baseline or day 1 (pre treatment). In the week number 4 (post treatment). Up to 8 weeks (follow-up). Through study completion, an average of 6 months.
  Questionnaire of 30 questions for quality of functional movement and 30 questions of quantity of functional movement of upper extremity. The maximal score is 150 for both quantity and quality.
Box and block test | It is administered in three stages: Baseline or day 1 (pre treatment). In the week number 4 (post treatment). Up to 8 weeks (follow-up). Through study completion, an average of 6 months.
  Patient must to pick up little boxes and carry on in a standarized box. Patient must perform the test with both hands, with paresis and without paresis in 1 minute per each upper extremity.
Medical research council | It is administered in three stages: Baseline or day 1 (pre treatment). In the week number 4 (post treatment). Up to 8 weeks (follow-up). Through study completion, an average of 6 months.
  Manual test muscle that use oxford graduation. M0 total weakness to M5 is normal strenght

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Alemana, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demeco A, Zola L, Frizziero A, Martini C, Palumbo A, Foresti R, Buccino G, Costantino C. Immersive Virtual Reality in Post-Stroke Rehabilitation: A Systematic Review. Sensors (Basel). 2023 Feb 3;23(3):1712. doi: 10.3390/s23031712. PMID 36772757
- [Derived] Peralta-Wieland B, Vasquez-Torres R, Maldonado-Diaz M, Yoma M. Immersive Virtual Reality-Based Rehabilitation for Upper Limb Recovery in Acute and Subacute Stroke Patients: A Feasibility Study. Physiother Res Int. 2026 Jan;31(1):e70151. doi: 10.1002/pri.70151. PMID 41416487